CLINICAL TRIAL: NCT03477136
Title: Correlation of Serum and Semen Vitamin D Level With Semen Parameters in Males
Brief Title: Serum and Semen Vitamin D Level With Semen Parameters
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mary Yonan, Principal investigator, Assiut University
Other Study IDs: SSVDSS
Record Dates: First submitted 2018-03-20; First posted 2018-03-26 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Semen Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples semen samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- First group: semen parameter showing normospermic: * group will include 30 male
  * Semen samples will be collected from all patients Semen analysis will be examined after 2-5 days of sexual abstinence based on World Health Organization (WHO) (2010)
  * blood and semen sample will be collected from all males to evaluate vitamin D level by ELISA .
  Interventions: Diagnostic Test: ELISA to evaluate serum and seminal vitamin D level
- second group: semen parameter asthenozoospermic: * group will include 30 male
  * Semen samples will be collected from all patients Semen analysis will be examined after 2-5 days of sexual abstinence based on World Health Organization (WHO) (2010)
  * blood and semen sample will be collected from all males to evaluate vitamin D level by ELISA .
  Interventions: Diagnostic Test: ELISA to evaluate serum and seminal vitamin D level
- Third group: semen parameter oligozoospermic: * group will include 30 male
  * Semen samples will be collected from all patients Semen analysis will be examined after 2-5 days of sexual abstinence based on World Health Organization (WHO) (2010)
  * blood and semen sample will be collected from all males to evaluate vitamin D level by ELISA .
  Interventions: Diagnostic Test: ELISA to evaluate serum and seminal vitamin D level
- Forth groupsemen parameter: astheno-teratozoospermic,: * group will include 30 male
  * Semen samples will be collected from all patients Semen analysis will be examined after 2-5 days of sexual abstinence based on World Health Organization (WHO) (2010)
  * blood and semen sample will be collected from all males to evaluate vitamin D level by ELISA .
  Interventions: Diagnostic Test: ELISA to evaluate serum and seminal vitamin D level
- Fifth group semen parameter: oligo asthenoteratozoospermia: * group will include 30 male
  * Semen samples will be collected from all patients Semen analysis will be examined after 2-5 days of sexual abstinence based on World Health Organization (WHO) (2010)
  * blood and semen sample will be collected from all males to evaluate vitamin D level by ELISA .
  Interventions: Diagnostic Test: ELISA to evaluate serum and seminal vitamin D level

INTERVENTIONS:
Diagnostic Test: ELISA to evaluate serum and seminal vitamin D level — Serum and semen samples will be collected from all participant males and ELISA method used to evaluate the level of vitamin D in serum and semen
  Other Names: semen analysis

SUMMARY:
vitamin D may have multiple functions, one of them is modulating reproductive processes and the reproductive role of vitamin D is highlighted by expression of the vitamin D receptors in testis, male reproductive tract and sperms

DETAILED DESCRIPTION:
Semen analysis is the corner stone of infertility evaluation as it provides information on the functional status of the seminiferous tubules, epididymis and accessory sex glands. The methods on how the semen should be evaluated are provided by the World Health Organization Vitamin D is synthesized mainly in the skin, where ultraviolet ray B radiation converts 7-dehydrocholesterol to Vitamin D3. Then, Vitamin D3 undergoes two hydroxylation processes first in the liver and second in the kidney Serum 25(OH)D is the major circulating metabolite of vitamin D and reflects vitamin D inputs from cutaneous synthesis and dietary intake. The serum 25(OH)D level is the standard clinical measure of vitamin D status Vitamin D deficiency has been linked to various health disorders including boneheallth, cardiovascular, infectious, oncologic, musculoskeletal, neuropsychologic and reproductive disorders, as well as to overall mortality

ELIGIBILITY:
Inclusion Criteria

* -males with different semen parameter finding
* Age: 20-50 years

Exclusion Criteria:

1. Varicocele.
2. Genital tract infections.
3. Primary and secondary hypogonadism
4. Hormonal therapy.
5. Calcium and vitamin D supplement.
6. Hepatic or renal failure
7. Diseases or drugs affecting vitamin D absorption -

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The patients will be recruited from the out patient clinic of Andrology, Assuit university hospital.
  One hundred and fifty individuals will be included divided into five groups according to semen parameters finding
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
correlation of serum and semen vitamin D level with semen parameters in males | A year
  evaluation the level of vitamin D in serum and semen by using ELISA method and correlate it with semen parameters

CONTACTS AND LOCATIONS:
Overall Officials: Mary Younan, Resident, Principal Investigator — Assiut Univeristy
Locations (1):
- Faculty of Medicine, Asyut, Egypt

REFERENCES:
- [Background] Blomberg Jensen M, Jorgensen A, Nielsen JE, Bjerrum PJ, Skalkam M, Petersen JH, Egeberg DL, Bangsboll S, Andersen AN, Skakkebaek NE, Juul A, Rajpert-De Meyts E, Dissing S, Leffers H, Jorgensen N. Expression of the vitamin D metabolizing enzyme CYP24A1 at the annulus of human spermatozoa may serve as a novel marker of semen quality. Int J Androl. 2012 Aug;35(4):499-510. doi: 10.1111/j.1365-2605.2012.01256.x. Epub 2012 Mar 9. PMID 22404291
- [Background] Esteves SC. Clinical relevance of routine semen analysis and controversies surrounding the 2010 World Health Organization criteria for semen examination. Int Braz J Urol. 2014 Jul-Aug;40(4):443-53. doi: 10.1590/S1677-5538.IBJU.2014.04.02. PMID 25254609
- [Background] Hammoud AO, Meikle AW, Peterson CM, Stanford J, Gibson M, Carrell DT. Association of 25-hydroxy-vitamin D levels with semen and hormonal parameters. Asian J Androl. 2012 Nov;14(6):855-9. doi: 10.1038/aja.2012.77. Epub 2012 Oct 8. PMID 23042450
- [Background] Herrmann M, Farrell CL, Pusceddu I, Fabregat-Cabello N, Cavalier E. Assessment of vitamin D status - a changing landscape. Clin Chem Lab Med. 2017 Jan 1;55(1):3-26. doi: 10.1515/cclm-2016-0264. PMID 27362963
- [Background] Yan WJ, Yu N, Yin TL, Liu L, Yang J. Can Vitamin D supplementation be used as adjunctive treatment for oligozoospermia or asthenozoospermia accompanied with Vitamin D deficiency? Asian J Androl. 2015 Jan-Feb;17(1):165-7. doi: 10.4103/1008-682X.138190. No abstract available. PMID 25219916